CLINICAL TRIAL: NCT06738329
Title: Investigating the Impact of the Seaweed Derived Food Additive, Carrageenan, on the Human Gut Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Cargill R&D Centre Europe, Havenstraat 84, 1800 Vilvoorde, Belgium (Unknown)
Responsible Party: Principal Investigator, Hannah Thomas, Miss, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: UREC24/21
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Gut Microbiome; Healthy Donors
Keywords: Carrageenan; Gut microbiome; Gut health; food additive
MeSH Terms: interventions — Carrageenan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Carrageenan gummy (Experimental): Gummies have been produced using carrageenan as a gelling agent. Each dose will consist of two carrageenan containing gummies
  Interventions: Other: Carrageenan gummy sweet
- Prebiotic arm (Experimental): The prebiotic fibre, inulin, has been added into the carrageenan gummies. Each dose with consist of two gummy sweets.
  Interventions: Other: Carrageenan and inulin gummy sweet
- Placebo (Placebo Comparator): An alternative gelling agent, agar has been added to the gummy sweets as a placebo.
  Interventions: Other: Placebo agar agar gummy

INTERVENTIONS:
Other: Carrageenan gummy sweet — Gummy sweet containing carrageenan and agar as the gelling agents.
  Arms: Carrageenan gummy
Other: Carrageenan and inulin gummy sweet — Gummy sweet containing agar and carrageenan as gelling agents, with added inulin.
  Arms: Prebiotic arm
Other: Placebo agar agar gummy — Gummy sweet containing agar as gelling agents.
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate whether a seaweed derived food additive, carrageenan, has an impact on the human gut microbiome in vivo. The primary purpose is to assess whether consumption of a carrageenan containing product for 4 weeks can alter the bacterial composition of the gut microbiome in healthy individuals and whether the addition of a prebiotic fibre, inulin, to the product has an enhanced beneficial impact of the gut composition. The main questions to answer are:

Does the consumption of a confectionary item containing carrageenan and inulin lead to a positive impact on the faecal microbial community when compared to the confectionary item containing no carrageenan and no inulin (placebo)? Participants will be asked to consume 2 gummy sweets for 4 week period and provide stool and urine samples on 3 occasions over a 9 week period.

Does the consumption of a confectionary item containing carrageenan and inulin improve gastrointestinal comfort measured using overall SHS-GI score when compared to baseline measurements recorded during run in period?

DETAILED DESCRIPTION:
Carrageenan is a frequently used food additive within the food industry. It acts as a gelling agent and thickener and is often used as a vegan alternative to gelatine. You will often see it on food labels as E407 or E407a. As a type of carbohydrate resistant to human digestion, the question has been posed as to whether carrageenan can be utilised by the gut microbiota (the community of microorganisms residing in the human gut). As the confectionary market remains a big part of daily life for many, having sweets that have a positive impact on the gut microbiota could be a step forward in promoting healthier snack choices. We have conducted lab-based experiments which have shown that carrageenan can be used by a number of gut microbial species, both beneficial and undesirable. We ascertained that consumption of carrageenan in low amounts in conjunction with prebiotics (dietary substrates selectively utilised by beneficial gut microorganisms which have a health benefit) can mitigate the growth of undesirable microbes, and overall have an enhanced beneficial effect on the microbial composition by promoting the growth on beneficial gut bacteria. This study aims to assess if these positive microbial changes can also be observed in humans, by conducting a human trial. We will adopt a randomised, double-blind parallel study design in which participants are either given 1) a carrageenan (0.167g) containing confectionary item 2) a carrageenan and inulin (5g) containing confectionary item or 3) a confectionary item containing an alternative gelling agent (control) to consume daily for 4 weeks. The dosage of carrageenan is comparable to what is found in commercially available sweets. The dosage of inulin is comparable to what previous studies found had a positive impact on the gut microbiome. Participants will be screened for eligibility prior to the study and given time to consider their participation. Once consent has been gained, participants will be asked to complete a 24 hour recall on 3 days during a 1 week run-in period (period prior to consuming the intervention/placebo). Participants will be asked to donate a stool and urine sample on the first day of the study. They will be asked to complete a Bristol stool chart daily (to monitor bowel habits) and a Short Health Scale for GastroIntestinal symptoms (SHS-GI) questionnaire daily (to monitor gastrointestinal symptoms) and to complete a second 3 -day dietary recall at the end of the 4 week intervention. On the last day of the 4 week intervention participants will be asked to give a second stool and urine sample. The participants will also be asked to give a third sample after a 4 week washout period (a period where participants will not consume any intervention). The purpose of this washout period it to assess whether any changes to the gut microbiota are reversed after 4 weeks. The collected stool and urine samples will be analysed using microbial and metabolic profiling to identify differences in gut microbiota composition and function. Participants will be allocated unique ID codes and will be given the opportunity to withdraw at any time during the study without explanation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Prescribed antibiotics in the last 3 months
* Individuals with any gut disorders such as IBS or IBD
* individuals with any food allergies or intolerances
* Individuals who regularly consume pre or probiotics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessing changes in microbial community post consumption of a carrageenan-inulin gummy. | 4 week intervention period
  Does the consumption of a confectionary item containing carrageenan and inulin lead to a positive impact on the faecal microbial community when compared to the confectionary item containing no carrageenan and no inulin (placebo)?

SECONDARY OUTCOMES:
Assessing changes in gastrointestinal comfort post carrageenan-inulin consumption | 4 week intervention period
  Does the consumption of a confectionary item containing carrageenan and inulin improve gastrointestinal comfort measured using overall SHS-GI score when compared to baseline measurements recorded during run in period?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided